CLINICAL TRIAL: NCT07220395
Title: Spanish Language Older Adult eHealth Learning
Brief Title: eHealth Literacy Intervention for Spanish Speaking Older Adults in the US
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 025-417; K01AG081455 (NIH)
Record Dates: First submitted 2025-10-18; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: eHealth Literacy
Keywords: Spanish speakers; eHealth; older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eHealth Training Group (Experimental): 4-week, twice a week eHealth literacy training intervention
  Interventions: Behavioral: eHiLLs

INTERVENTIONS:
Behavioral: eHiLLs — Adapted intervention for Spanish speaking older adults.

SUMMARY:
The PI will assess the feasibility and acceptability of an eHealth literacy intervention with Spanish-preferred older adult Latinos. This proposal will generate novel data to justify a future R01 proposal to advance aging research with high-risk populations and assess the efficacy of the intervention.

DETAILED DESCRIPTION:
C. Approach C.1 Overview. In aim 3, the PI will assess the feasibility and acceptability of the intervention with Spanish-preferred older adult Latinos. Combined with a rigorous training plan, working with top experts in the fields of aging, Latino health, implementation science, and technology-based intervention development, this proposal will generate novel data to justify a future R01 proposal to advance aging research with underrepresented populations and assess efficacy with a larger sample.

C.2 Changes in Design. Previous versions of the intervention have been guided by the literature on older adults' learning of computer technology, and feature key elements designed specifically to accommodate older computer learners' needs and preferences. These include (1) providing step-by-step, detailed instructions and avoiding technical jargon, (2) providing hands-on practice and encouraging questions, (3) making sure each lesson builds on previous lessons and increases complexity gradually, (4) ensuring the learners experience at least some level of success at the initial stage of the training6, (5) conducting the training in a familiar, relaxed, and supportive environment, and (6) offering the training in the early morning hours, which is generally the optimal time of day for older learners. These elements remain key components of the intervention.

These changes have been made for two reasons. First, due to changes in people's way of living post-COVID (i.e., less in-person contact), in-person intervention delivery may not be acceptable as a delivery method for older adults who continue to be a vulnerable group as COVID shifts from a pandemic to an endemic. Additionally, interaction with healthcare systems is increasingly moving online. Thus, virtual learning with a live facilitator synchronously over Zoom may be a more acceptable approach. Second, the literature assessing interventions with Latino populations suggests the use of peer advisors (i.e., promotoras or Lay-health Advisors) has emerged as a potentially effective approach for improving access to care, health outcomes, and health behaviors. Wisniewski et al. proposed the importance of a new role in healthcare, in which peers assist others in navigating technology to take advantage of new tools that augment existing pathways to good health and healthcare. The emergence of the use of peer advisors (promotoras) is a natural progression for healthcare as the role of technology expands, so will the need to support its implementation. The next section describes the cultural adaptation process and further justifies the need of a peer advisor (promotora) in intervention work with Latino populations.

C.3 Cultural Adaptation. In addition to including promotoras and having the intervention materials translated into Spanish, cultural adaptation goes beyond language to focus on factors relevant to the Latino community. The literature provides practical steps for culturally adapting interventions for adult Latinos. Much of the literature in this area comes from one of the mentors on this proposal, as a pioneer in cultural adaption with Latino populations and internet-based interventions

Religion. Muñoz and Mendelson suggest incorporating religion, particularly Catholicism, often resonates with Latino participants who use religion as an important lens when making decisions. The use of relevant phrases or "dichos" to motivate and engage participants is another important part of cultural adaptation and this can be paired with incorporation of religion. For example, Latinos often use the phrase "si Dios quiere" ("what God wants"), which can guide their perception about control over aspects of their health. Subjects' beliefs can be used as a counter to what subjects perceive as barriers. For example, suggesting God brought this intervention into their lives and addressing the concept that God helps those who help themselves.

Family. Another factor that can be used for motivation in the intervention is emphasizing family or familismo. Familismo is an important part of health decision-making as close friends and family are often consulted before medical professionals. This can be used as a motivating factor by reinforcing that learning eHealth will help their family, such as suggesting that subjects will be able to share this knowledge (i.e., help their husband) or explaining how this could lead to good health to help them live longer and be around family longer.

Respect. It is important to select resources and strategies that provide a balance between one's culture of origin and the culture in which subjects now live. This helps establish respect of one's culture of origin and enhance self-efficacy by reducing the burden of learning all new resources and strategies from the dominant culture. Muñoz and Mendelson found that one way to help Latinos learn new strategies is to provide a peer facilitator that shares a familiar background and language. This also helps acknowledge lived experiences because a peer facilitator may allow participants to feel safe to discuss issues that affect how subjects interact with healthcare systems. Another strategy to consider is the use of formal titles with older adults as a sign of respect.

Latino Heterogeneity. A major consideration when working with Latino populations is that different Latino subgroups may respond differently as there is variability across these subgroups. For example, Mexican might use the term "listo" to mean 'ready' whereas El Salvadorans may use the term "aguja" to mean the same thing. Acknowledging not all Latinos share the same lived experiences is critical to respecting the variability within the U.S.-based Latino population. Assessing how Latinos from different subgroups respond to the adaptations will be important for future research. The PI will be intentional during recruitment to consider Latinos from various countries and experiences.

Throughout the adaptation process, the PI will receive feedback from mentors on the project and from a Community Advisory Board. The Community Advisory Board will comprise stakeholders from the partnerships mentioned in section

C.4 Assessing Feasibility and Acceptability of Culturally Adapted Intervention. The importance of conducting preliminary studies prior to implementation of interventions is well documented. It is important to define the purpose a feasibility and acceptability study to explain how this is not an efficacy study. The primary role of a feasibility study is to test all aspects of a research protocol and ensure the procedures work as desired. The study will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework. RE-AIM provides a practical means of evaluating behavioral health change interventions. Using RE-AIM, the impact of innovations can be assessed at both the individual (i.e., end-user) and organizational (i.e., delivery agent) levels. The proposed work will answer questions in preparation for the implementation of a fully powered study, such as: How were participants recruited? Was recruitment successful? What percent of people contacted agreed to participate? What percent of people who agreed actually participated? Were all baseline participants retained for post assessments? Why was there dropout? What were the characteristics of those retained in the sample versus those lost (i.e., retention bias)? Were the investigators able to deliver the intervention? As intended (i.e., fidelity)? Did participants do what the team wanted? Did the subjects face problems in doing it? Were the investigators able to implement our measures pre and post? Were the scales the investigators employed shown to be reliable in this sample? With this information, a fully powered study with fewer problems will be implemented to test the efficacy. Questions related to whether the recruitment, intervention delivery, facilitators, activities, and outcome measures were acceptable will be asked to assess acceptability and satisfaction from participants. The proposed research is not assessing efficacy and will answer the questions above and more to assess feasibility and acceptability for a larger study. Table 3 provides examples of the primary objectives, based on the questions above and prior studies, and how those objectives will be measured. All mentors have successfully conducted feasibility studies to guide the PI during this work.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older,
* Spanish is preferred language,
* are of Latino descent,
* are physically able to use computer or mobile device (i.e., tablet)

Exclusion Criteria:

* Major cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
eHealth Literacy Scale | From enrollment to end of intervention at 4 weeks.
  Measures the degree to which individuals have the capacity to obtain, process, and understand basic health information and services needed to make appropriate health decisions. 8-item measure.
  The scale is 0 to 8. Higher score mean better eHealth literacy.
  Norman CD, Skinner HA. eHealth literacy: essential skills for consumer health in a networked world. Journal of Medical Internet Research. 2006 Jun 16;8(2):e506.

IPD SHARING:
Plan to Share IPD: No